CLINICAL TRIAL: NCT00168311
Title: A Double-Blind Placebo Controlled Trial of Repetitive Transcranial Magentic Stimulation (rTMS) in the Treatment of Negative Symptoms in Schizophrenia and Related Disorders
Brief Title: A Double-Blind Placebo Controlled Trial of Repetitive Transcranial Magnetic Stimulation (rTMS) in the Treatment of Negative Symptoms in Schizophrenia
Acronym: rTMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Alfred (Other)
Responsible Party: Principal Investigator, Assoc Professor Paul Fitzgerald, Professor, The Alfred
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 81/02
Record Dates: First submitted 2005-09-14; First posted 2005-09-15 (Estimated); Results first posted 2012-05-14 (Estimated); Last update posted 2012-05-14 (Estimated); Status verified 2012-04

CONDITIONS: Schizophrenia
Keywords: Transcranial Magnetic Stimulation; Schizophrenia; Negative Symptoms
MeSH Terms: conditions — Schizophrenia | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Treatment (Experimental): Bilateral high frequency (10 Hertz) rTMS
  Interventions: Device: Transcranial Magnetic Stimulation
- Sham rTMS (Sham Comparator): Bilateral Sham rTMS
  Interventions: Device: sham TMS

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — Participants were sequentially randomly assigned to either 15 active bilateral treatments or 15 sham bilateral treatments that were administered on a daily basis, five days per week.
  Arms: Active Treatment
Device: sham TMS
  Arms: Sham rTMS

SUMMARY:
There is pilot data to suggest the therapeutic value of rTMS applied to the left prefrontal cortex in the treatment of negative symptoms. Neuroimaging studies demonstrate abnormal activity in this region in patients experiencing negative symptoms. Finally rTMS applied at high frequency shows the capacity to up-regulate cortical activity in a way that would provide an explanation for a therapeutic response.

The study involves participants receiving 15 sessions of high frequency rTMS treatment applied bilaterally to the prefrontal cortex over a 3 week period or sham rTMS. Following this double blind phase, participants randomised to placebo treatment will be offered 15 sessions of active treatment.

In addition, ppTMS (paired pulse TMS) will be conducted prior to the onset of treatment and after completion of the course, as a means of measuring cortical inhibition and facilitation. NIRS (Near Infra red spectroscopy) will also be conducted prior to, during and after the first and last treatment sessions to allow monitoring of oxygenated and deoxygenated haemoglobin.

DETAILED DESCRIPTION:
The main outcome measure used is the SANS (Scale for the Assessment of Negative Symptoms. This is a semi strucutured interview which provides scores from 0-70. This is administered at baseline, week 2, 3, 5 and 6.

Other outcome measures administered are (frequency mentioned above): PANSS (Positive and Negative Syndrome Scale) and the Calgery Depression Scale for Schizophrenia, A cognitive battery is also administered.

Inclusion Criteria:

* Diagnostic and Statistical Manual-IV diagnosis of schizophrenia or schizoaffective disorder, age over 18
* Persistent negative symptoms of moderate to severe intensity
* Failure to respond to a minimum of two antipsychotic medications
* No increase or initiation of new antipsychotic therapy in the four weeks prior to entering the trial Exclusion Criteria
* Prominent positive symptoms
* Have an unstable medical condition, neurological disorder or any history of seizure disorder or are currently pregnant or lactating
* Previous brain injury or surgery, any metal clips, plates or other metal items in the head, cardiac pacemaker
* Subjects at high risk of violence or suicide as determined by the investigator and treating clinicians
* Substance dependence

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of schizophrenia or schizoaffective disorder, age over 18
* Persistent negative symptoms of moderate to severe intensity
* Failure to respond to a minimum of two antipsychotic medications
* No increase or initiation of new antipsychotic therapy in the four weeks prior to entering the trial

Exclusion Criteria:

* Prominent positive symptoms
* Have an unstable medical condition, neurological disorder or any history of seizure disorder or are currently pregnant or lactating
* Previous brain injury or surgery, any metal clips, plates or other metal items in the head, cardiac pacemaker
* Subjects at high risk of violence or suicide as determined by the investigator and treating clinicians
* Substance dependence

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2002-08; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul B Fitzgerald, MBBS, PhD, Principal Investigator — Alfred Psychiatry Research Centre
Locations (1):
- Alfred Psychiatry Research Centre, Melbourne, Victoria, Australia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 20 patients were randomly assigned. Patients were recruited from the outpatient department of two public area mental health services and by referral from a number of private psychiatrists between January 2003 and July 2007.
Groups:
- Active Treatment: Bilateral high frequency (10Hz) rTMS
- Sham Treatment: Sham bilateral rTMS treatment
Period: Overall Study
Arm/Group | Active Treatment | Sham Treatment
Started | 12 | 10
Completed | 12 | 8
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Treatment | Sham Treatment | Total
Number analyzed (Participants) | 12 | 10 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 10 | 22
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — 16 men and 4 women
  Participants
    Female | 2 | 2 | 4
    Male | 10 | 8 | 18
Region of Enrollment [Number; unit: participants]
  Australia | 12 | 10 | 22

OUTCOME MEASURES:

1. Primary Outcome: Scale for the Asessment of Negative Symptoms (SANS)
Description: Scale for Assessment of Negative Symptoms [SANS]. This is a semi structured interview. Assessments are conducted on a six-point scale (0=not at all to 5=severe)with a total score range of 0-70. A score of >50 is considered to be a moderate-severe intensity.
Time Frame: 3 weeks
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Active Treatment | Sham Treatment
Number analyzed (Participants) | 12 | 8
Scores on a scale | 38.8 (11.0) | 53.7 (8.3)

ADVERSE EVENTS:
Arm/Group | Active Treatment | Sham Treatment
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/10
Other Adverse Events (participants affected / at risk) | 0/12 | 0/10

LIMITATIONS AND CAVEATS:
Insufficient time period used to be able to establish a substantive therapeutic effect of rTMS; standard dosing method may be inadequate due to volumetric changes in brain regions in schizophrenia; concurrent antipsychotic medication.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No